CLINICAL TRIAL: NCT05105100
Title: Peripheral T Cell Determinants of Response and Resistance to Pembrolizumab in Melanoma
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 21853
Record Dates: First submitted 2021-10-12; First posted 2021-11-03 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Melanoma; Advanced Melanoma
Keywords: Peripheral T Cell; Pembrolizumab
MeSH Terms: conditions — Melanoma | interventions — Biopsy; Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Melanoma: Participants will undergo a pre-treatment tumor core biopsy and Peripheral blood mononuclear cell (PBMC) collection. Then, patients will be started on pembrolizumab per standard of care and PBMCs will be collected every 3 weeks (1 cycle)
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biopsy — Tumor tissue collection
  Other Names: Excisional Biopsy
Procedure: Biospecimen Collection — Intravenously Blood draw
  Other Names: Specimen Collection

SUMMARY:
This is a non-therapeutic study assessing peripheral T cell determinants of response and resistance to immunotherapy in patients with advanced melanoma.The hypothesis is that systemic T cells traffic into the tumor microenvironment (TME) can predict response and resistance to immunotherapy. These systemic tumor directed T cells can be defined by tumor/blood small conditional RNA (scRNA) using T cell receptor (TCR) as a barcode and can help predict response to PD-1 therapy.

DETAILED DESCRIPTION:
Primary Objective:

To understand how the systemic immune profile (T cell activation and expansion in TME) changes in response to pembrolizumab therapy in patients with advanced melanoma on pembrolizumab monotherapy.

Exploratory Objectives :

I. To correlate the peripheral T cell profiles with the objective response rate (ORR) at 24 weeks in patients with advanced melanoma on pembrolizumab monotherapy.

II. To correlate the peripheral T cell profiles with progression free survival (PFS) in patients with advanced melanoma on pembrolizumab monotherapy.

III. To correlate the peripheral T cell profiles with overall survival (OS) in patients with advanced melanoma on pembrolizumab monotherapy.

IV. To correlate the peripheral T cell profiles with toxicity profile. V. Transcriptional and phenotypic features of tumor directed T cells in blood using a combination of phenotypic markers derived from COMET and cite-seq.

Patients will be followed for 6 months from time of treatment initiation. After 6 months, patients do not need to be followed but standard of care scans and survival status can be assessed for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed locally advanced or metastatic melanoma and be starting on standard of care pembrolizumab monotherapy. Patients may have received any or no prior anti-cancer therapy without limitation.
2. Must have one or more sites of disease amenable to biopsy (tumor, skin, lymph node, pleural fluid, peritoneal fluid, cerebral spinal fluid (CSF)).
3. Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
4. Participants must be age 18 years or older on the day of signing informed consent.
5. Have the ability to provide written informed consent for the trial.
6. Be able and willing to comply with study procedures including provision of basic demographic information and medical history.
7. Be willing to receive periodic follow up phone calls to monitor health status and survival status.

Exclusion Criteria:

1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX 40, Cluster of Differentiation 137 (CD137)).
2. Has received prior systemic anti-cancer therapy including investigational agents within the prior 2 weeks.
3. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
4. Has a contraindication to tissue biopsy for minimally-invasive research-procedure
5. Contraindication to phlebotomy (up to 20 milliliters (mL)) per phlebotomy every three weeks).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Melanoma and Cutaneous Oncology Program at the Helen Diller Family Comprehensive Cancer Center at University of California San Francisco.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Number of genes predictive of response at Baseline | Baseline
  The investigators will identify the genes predictive of response to anti-PD-1 therapy by testing for significant associations across expression rates of each gene and response/resistance, within a hurdle-Gaussian mixed-effect framework that accounts for variance across patients and technical noise present in single-cell data.
Number of genes predictive of response at 24 weeks | 24 weeks
  The investigators will identify the genes predictive of response to anti-PD-1 therapy by testing for significant associations across expression rates of each gene and response/resistance, within a hurdle-Gaussian mixed-effect framework that accounts for variance across patients and technical noise present in single-cell data.
Number of T-cell sub-populations | Baseline and 24 weeks
  The investigators will identify T cell sub-populations in the tumor-directed component in blood whose relative frequency is indicative of response to anti-PD-1 therapy, using a negative binomial regression model. We will test for predictive differences in relative frequencies before and after treatment initiation separately, as well as when combining both time points with appropriate interaction terms
Proportion of participants with a change in clonal expansion of T cells associated with response to anti-PD-1 therapy | 24 weeks
  The investigators will build a novel computational framework to identify T-cell clonal behavior associated with response to anti-PD-1 therapy using profiling of TCR sequences at single-cell resolution to compare clonal expansion in each of the sub-populations for their association with response to anti-PD-1 therapy.
Proportion of participants with a change in distribution of T cells associated with response to anti-PD-1 therapy | 24 weeks
  The investigators will build a novel computational framework to identify T-cell clonal behavior associated with response to anti-PD-1 therapy using profiling of TCR sequences at single-cell resolution to compare distribution of T cells in each of the sub-populations for their association with response to anti-PD-1 therapy.
Number of transcriptional migration events | 24 weeks
  The investigators will search for "transcriptional migration" events, in which T cell clones change their transcriptional profile following treatment and will assess the predictive power of such events to the success of anti-PD-1 therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Adil Daud, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No